CLINICAL TRIAL: NCT01151943
Title: Comparison of Two Methods of Pain Relief After Cesarean Delivery: Transversus Abdominis Plane (TAP) Block Versus Incisional Infiltration With Local Anesthetic
Brief Title: Comparison of Two Types of Pain Relief After Cesarean Delivery
Acronym: Cesar-Dol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been halted prematurely beacuse of the occurence of convulsions in one case after TAP block.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/15; 2010-019662-88 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Cesarean Section
Keywords: cesarean section; continuous wound infiltration; transversus abdominis plane block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transversus Abdominis Plane (TAP) Block (Experimental): Patients will receive a bilateral transversus abdominis plane block
  Interventions: Other: Transversus Abdominis Plane (TAP) Block
- Incisional Infiltration of Local Anesthetic (Active Comparator): Patients will receive an incisional infiltration with local anesthetic (continuous administration of levobupivacaïne during 48 hours)
  Interventions: Other: Incisional Infiltration of Local Anesthetic

INTERVENTIONS:
Other: Transversus Abdominis Plane (TAP) Block — Bilateral injection of levobupivacaine (20 mL, 3.75 mg/mL)
  Arms: Transversus Abdominis Plane (TAP) Block
Other: Incisional Infiltration of Local Anesthetic — continuous administration of levobupivacaine (1,25 mg/mL,5 mL/h) during 48 hours.
  Arms: Incisional Infiltration of Local Anesthetic

SUMMARY:
Women undergoing elective cesarean delivery, performed under a standard spinal anesthesia, will be randomized to undergo either TAP block or incisional infiltration with local anesthetic, in addition to standard postoperative analgesia comprising regular acetaminophen, nefopam and ketoprofen. Short acting oral morphine will be given as a rescue treatment in case of severe pain.

ELIGIBILITY:
Inclusion Criteria:

* scheduled cesarean section performed under spinal anesthesia
* ASA I or II
* height above 1,55 m
* singleton pregnancy

Exclusion Criteria:

* contre indication to a drug used in the study (levobupivacaine, ketoprofen, nefopam)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
severity of postoperative pain | 48 postoperative hours

SECONDARY OUTCOMES:
delay before the first rescue dose of morphine | 48 postoperative hours
morphine requirement | 48 postoperative hours
complication of each loco-regional technique | end of hospitalisation
patient's satisfaction | end of hospitalisation
length of hospital stay | end of hospitalisation
occurrence of a neuropathic postoperative pain | 1 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

REFERENCES:
- [Derived] Chandon M, Bonnet A, Burg Y, Barnichon C, DesMesnards-Smaja V, Sitbon B, Foiret C, Dreyfus JF, Rahmani J, Laloe PA, Fischler M, Le Guen M. Ultrasound-guided Transversus Abdominis plane block versus continuous wound infusion for post-caesarean analgesia: a randomized trial. PLoS One. 2014 Aug 5;9(8):e103971. doi: 10.1371/journal.pone.0103971. eCollection 2014. PMID 25093663